CLINICAL TRIAL: NCT03891862
Title: A Phase 4, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Evaluate the Persistence of Effect and Safety of Valbenazine for the Treatment of Tardive Dyskinesia
Brief Title: Persistence of Effect and Safety of Valbenazine for the Treatment of Tardive Dyskinesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NBI-98854-TD4002
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Tardive Dyskinesia (TD)
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-label Valbenazine (Experimental): Participants received valbenazine 40 mg once daily for 1 week, then 80 mg once daily for the remainder of the 8-week open label period.
  Interventions: Drug: Valbenazine
- Placebo-controlled Placebo (Placebo Comparator): Participants received placebo (matching valbenazine) once daily for 8 weeks. Randomization into this arm occurred after open-label treatment with valbenazine once daily for 8 weeks.
  Interventions: Drug: Placebo oral capsule
- Placebo-controlled Valbenazine (Experimental): Participants received valbenazine 80 mg once daily for 8 weeks. Randomization into this arm occurred after open-label treatment with valbenazine once daily for 8 weeks.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — vesicular monoamine transporter 2 (VMAT2) inhibitor
  Other Names: Ingrezza, NBI-98854
  Arms: Open-label Valbenazine; Placebo-controlled Valbenazine
Drug: Placebo oral capsule — non-active dosage form
  Arms: Placebo-controlled Placebo

SUMMARY:
This is a Phase 4, randomized, double-blind, placebo-controlled study to evaluate the persistence of effect of valbenazine 40 mg and 80 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of childbearing potential must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment, and follow-up periods of the study.
2. Have one of the following clinical diagnoses for at least 3 months before screening: Schizophrenia, Schizoaffective Disorder, or Mood Disorder
3. Have a clinical diagnosis of neuroleptic-induced TD for at least 3 months before screening.
4. Be on stable doses if using maintenance medication(s) for schizophrenia or schizoaffective disorder, or mood disorder. Subjects with bipolar disorder must be on stable doses of a mood stabilizer.
5. Be in general good health.
6. Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month before screening.
2. Have a known history of substance (drug) dependence, or substance or alcohol abuse.
3. Have a significant risk of suicidal or violent behavior.
4. Have been hospitalized for psychiatric disorder within 6 months before Day 1.
5. Have a known history of neuroleptic malignant syndrome.
6. Have a known history of long QT syndrome or cardiac arrhythmia.
7. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed).
8. Are currently taking tetrabenazine or deutetrabenazine, or have used valbenazine (INGREZA) within 30 days of screening.
9. Have received an investigational drug within 30 days before Day 1 or plan to use an investigational drug (other than NBI-98854) during the study.
10. Have a blood loss ≥550 mL or donated blood within 30 days prior to Baseline.
11. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors (eg, tetrabenazine, deutetrabenazine).
12. Are currently pregnant or breastfeeding.
13. Have HIV or hepatitis B.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Chief Medical Officer
Locations (39):
- United States (38):
  - Neurocrine Clinical Site, Little Rock, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Costa Mesa, California
  - Neurocrine Clinical Site, Escondido, California
  - Neurocrine Clinical Site, Fountain Valley, California
  - Neurocrine Clinical Site, Glendale, California
  - Neurocrine Clinical Site, La Habra, California
  - Neurocrine Clinical Site, Lemon Grove, California
  - Neurocrine Clinical Site, Norwalk, California
  - Neurocrine Clinical Site, San Bernardino, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Pueblo, Colorado
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, North Miami, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, South Bend, Indiana
  - Neurocrine Clinical Site, Bloomfield Hills, Michigan
  - Neurocrine Clinical Site, East Lansing, Michigan
  - Neurocrine Clinical Site, Grand Rapids, Michigan
  - Neurocrine Clinical Site, Kansas City, Missouri
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Las Vegas, Nevada
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, Beachwood, Ohio
  - Neurocrine Clinical Site, Mason, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Conshohocken, Pennsylvania
  - Neurocrine Clinical Site, Scranton, Pennsylvania
  - Neurocrine Clinical Site, Franklin, Tennessee
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Houston, Texas
  - Neurocrine Clinical Site, Irving, Texas
  - Neurocrine Clinical Site, Richmond, Texas
  - Neurocrine Clinical Site, Petersburg, Virginia
  - Neurocrine Clinical Site, Spokane, Washington
- Neurocrine Clinical Site, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled male and female participants, 18 to 85 years of age, from 28 centers in the United States. Participants must have clinical diagnoses of schizophrenia or schizoaffective disorder with neuroleptic-induced tardive dyskinesia (TD) or mood disorder with neuroleptic-induced TD and have moderate or severe TD as assessed by an external Abnormal Involuntary Movement Scale (AIMS) Reviewer. The first and last participant was enrolled on 18 March 2019 and 3 September 2019, respectively.
Pre-assignment Details: After receiving valbenazine 40 mg for the first week followed by valbenazine 80 mg for 7 weeks during the open-label period, participants were randomly assigned to either placebo or to continue to receive valbenazine 80 mg.
Period: Open-label Period
Arm/Group | Open-label Valbenazine | Placebo-controlled Placebo | Placebo-controlled Valbenazine
Started | 135 | 0 | 0
Safety Analysis Set (The safety analysis set for the open-label valbenazine group in this period includes all participants who received at least one dose of study drug and have any post-baseline safety data collected.) | 132 | 0 | 0
Completed | 119 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: Placebo-controlled Period and Follow-up
Arm/Group | Open-label Valbenazine | Placebo-controlled Placebo | Placebo-controlled Valbenazine
Started (One participant who completed the open-label period was not randomized.) | 0 | 59 | 59
Persistence of Effect Analysis Set (Persistence of Effect analysis set included all randomized participants who received at least one dose of randomized study drug and have at least one AIMS assessment during the placebo-controlled period.) | 0 | 58 | 59
Completed Placebo-controlled Period | 0 | 53 | 56
Completed | 0 | 53 | 55
Not Completed | 0 | 6 | 4
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Persistence of effect analysis set, which includes all randomized participants who received at least one dose of randomized study drug and have at least one AIMS assessment during the placebo-controlled period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-controlled Placebo | Placebo-controlled Valbenazine | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (8.3) | 58.0 (8.0) | 58.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 57
  Male | 31 | 29 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 32 | 64
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 16 | 37
  White | 36 | 43 | 79
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Abnormal Involuntary Movement Scale at Study Baseline [Mean (Standard Deviation); unit: Score on scale] — The Abnormal Involuntary Movement Scale (AIMS) rates 10 items of involuntary movement, each item ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Items assess facial, oral, extremity, and trunk movements, as well as self-awareness of abnormal movements. The AIMS Dyskinesia Total Score is the sum of items 1-7 and ranges from 0 to 28, with higher scores indicating more severe dyskinesia.
  Score on scale | 10.3 (3.7) | 11.0 (4.1) | 10.7 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization (Week 8) in Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score at Week 16
Description: The AIMS rates 10 items of involuntary movement, each item ranging from 0 (no dyskinesia) to 4 (severe dyskinesia). Items assess facial, oral, extremity, and trunk movements, as well as self-awareness of abnormal movements. The AIMS Dyskinesia Total Score is the sum of items 1-7 and ranges from 0 to 28, with higher scores indicating more severe dyskinesia. Least-squares mean were estimated using a mixed-effects model for repeated measures.
Time Frame: Week 8, Week 16
Population: Persistence of effect analysis set, which includes all randomized participants who received at least one dose of randomized study drug and have at least one AIMS assessment during the placebo-controlled period. Participants who do not have an AIMS assessment at a scheduled or mapped early termination visit are not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Placebo-controlled Placebo | Placebo-controlled Valbenazine
Number analyzed (Participants) | 56 | 58
Score on scale | 0.6 [-0.8 to 1.9] | -1.6 [-3.0 to -0.3]

2. Secondary Outcome: Change From Baseline in the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Health State Index Score at Week 16
Description: The EQ-5D-5L assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The health state index score is based on the results of the individual health profiles using the United States value set and ranges from -0.573 to 1.0, with higher scores indicating higher health utility.
Time Frame: Baseline, Week 16
Population: Includes all participants who received at least one dose of study drug and have at least one postbaseline assessment. Missing data were imputed with last observation carried forward.
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo-controlled Placebo | Placebo-controlled Valbenazine
Number analyzed (Participants) | 57 | 59
Score on scale | 0.09 (0.03) | 0.16 (0.03)

3. Secondary Outcome: Change From Baseline in the EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Visual Analogue Scale (VAS) at Week 16
Description: The EQ-5D-5L assesses general health-related quality of life. The second portion of the scale is a self-perceived health score assessed using a VAS that ranges from 0 ("the worst imaginable health") to 100 ("the best imaginable health").
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Placebo-controlled Placebo | Placebo-controlled Valbenazine
Number analyzed (Participants) | 57 | 59
Score on scale | 4.5 (2.5) | 6.5 (2.8)

ADVERSE EVENTS:
Time Frame: Open-label valbenazine group: from baseline up to randomization (Week 8). Placebo-controlled placebo and valbenazine groups: from randomization (Week 8) up to Week 20
Arm/Group | Open-label Valbenazine | Placebo-controlled Placebo | Placebo-controlled Valbenazine
All-Cause Mortality (participants affected / at risk) | 1/132 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 3/132 | 2/59 | 1/59
Other Adverse Events (participants affected / at risk) | 17/132 | 11/59 | 7/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Valbenazine (N=132) | Placebo-controlled Placebo (N=59) | Placebo-controlled Valbenazine (N=59)
Cellulitis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Valbenazine (N=132) | Placebo-controlled Placebo (N=59) | Placebo-controlled Valbenazine (N=59)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 4 | 6 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2
Blood glucose increased (Investigations) | 0 | 0 | 2
Weight increased (Investigations) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03891862/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT03891862/SAP_001.pdf